CLINICAL TRIAL: NCT02123680
Title: Non-specific Chronic Low Back Pain Patients' Expectations Toward Physiotherapy and Physiotherapists: An Interpretive Socio-anthropological Study on Ill Persons' Experience
Brief Title: Chronic Low Back Pain Patients' Expectations Toward Physiotherapy
Acronym: CLBPEXPECT
Status: Completed | Type: Observational
Sponsor: Haute Ecole de Santé Vaud (Other)
Collaborators: HES-SO Commission scientifique du domaine santé (Unknown)
Responsible Party: Sponsor
Other Study IDs: 55-O13; 38495 (Other: HES-SO)
Record Dates: First submitted 2014-04-11; First posted 2014-04-25 (Estimated); Last update posted 2015-06-03 (Estimated); Status verified 2015-06

CONDITIONS: Chronic Low Back Pain
Keywords: expectation; chronic illness; trajectory
MeSH Terms: conditions — Chronic Disease

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Non-specific chronic low back pain guidelines recommend rehabilitation along with a biopsychosocial approach. However, though psychological and social issues address important needs of professionals and patients, they have been scarcely developed in this area so far. Noteworthy, little is known about patients' expectations relative to physiotherapy for chronic low back pain (CLBP), while professional recommendations advocate taking them into consideration.

A study about patients' experience will provide knowledge about the ill person's perspective and how the physiotherapists are perceived as well as the role attributed to them. The aim of this study is, thus, to explore the experience of the patients suffering from CLBP in order to highlight their expectations toward physiotherapy services and physiotherapists.

The investigators will apply a critically interpretive socio-anthropological approach based on patients' interviews and observations in an intensive CLBP rehabilitation program. The results will help improve the care patients receive by facilitating the integration of biopsychosocial issues related to patient's expectations into the treatment.

DETAILED DESCRIPTION:
INTRODUCTION

Chronic low back pain (CLBP) is defined as "pain and discomfort, localised below the costal margin and above the inferior gluteal folds, with or without referred leg pain" persisting for at least 12 weeks. It is classified as non-specific when "not attributable to a recognisable, known specific pathology, disorder, radicular syndrome or cauda equina syndrome". It is a very frequent condition, one year prevalence being around 25% for men and 35% for women. It can greatly alter functional capacity and quality of life. Including care, sick leave and work loss, it accounts for most of the back pain related costs.

Recommended management of CLBP is multidisciplinary due to the biopsychosocial impact of this condition. Most guidelines include the patient's education, advice to stay active, anti-inflammatory and analgesic medication, exercise therapy, and spinal manipulation. Multidisciplinary rehabilitation, adjunctive analgesics, and cognitive behavioural therapy are recommended if the initial approach is not efficient. Self-management strategies, self-monitoring of status, and decision-making are also promoted.

Physiotherapy plays a role in CLBP management, in collaboration with other health and social professions. As defined by the World Confederation for Physical Therapy, "Physiotherapy provides services to individuals and populations to develop, maintain and restore maximum movement and functional ability throughout the lifespan. (…) Functional movement is central to what it means to be healthy (…).This encompasses physical, psychological, emotional, and social wellbeing

Local and international standards of physiotherapy practice advocate taking patients' expectations into consideration. Physiotherapists are also advised to take patients preferences into account, when applying evidence-based practice (EBP) guidelines. However, knowledge about the expectations of patients toward physiotherapy is limited.

This research is conducted with an interdisciplinary approach. Indeed, it takes into account both the physiotherapy and the anthropological discipline. Physiotherapists want to deepen their comprehension of the patients' needs in order to take better care of them whereas anthropologists are interested in the broader experience of chronic illness and in understanding the relationship between cares and patients. With their concepts and qualitative methods, the latter have relevant tools to answer the research question.

Expectations issues within the CLBP rehabilitation process

Commonly, expectations are understood as "a belief that someone will or should achieve something". In the health field literature, the notion of expectation is often used, although it is seldom defined. Nevertheless, three dimensions emerge from the literature on CLBP patients' expectations: effectiveness of care (diagnosis, effective treatment, pain relief), relational issues (understanding, partnership, be believed, be treated as a person), and empowerment (self-management, exercise, advice, explanation, etc). In addition, expectations appear to be influenced by the course, the prognosis and the outcome of the rehabilitation.

CLBP patients are often dissatisfied with back pain rehabilitation. As pain relief is slight, disappointment with outcome is frequent. Having a clear diagnosis is clearly expected. Thus, additional medical investigations are frequently requested to find a cause to the disease. The patients also have expectations with regard to the outcome. Health professionals are expected to demonstrate communication skills, understand emotional and physical impact, spend time with the patient, show respect and build a partnership. They are also expected to understand the personal situation, demonstrate empowering skills, and adapt their language.

The nature of CLBP thus puts health professionals in an uncomfortable position. The diagnostic uncertainty and the limited effect of therapy challenge their competencies. The professional recommendations advise to avoid complex investigations and to stay active despite the pain. This position may be difficult to have when the patient wishes to obtain a clear diagnosis or to be prescribed time to rest for example. Thus, unrecommended approaches are sometimes implemented to maintain the relationship with the patient.

Patients' expectations of a diagnosis and a cure are in line with a biomedical approach, while a biopsychosocial model applies to CLBP treatment. It requires subtle interaction to bring the patient to consider that psychosocial issues influence pain and disability without giving the impression that pain is "in the mind" or exaggerated. This is especially difficult in a context where the person feels delegitimized. Indeed, disbelief and delegitimization by health professionals are motives for dissatisfaction.

Unclear diagnosis and poor social recognition

In Social sciences, the few studies that have explored the experience of CLBP patients show that, since they face long term diagnostic uncertainty, this places them in a liminal state being both well and sick, and being neither. Struggling for a diagnosis is an important source of strain added to the experience of pain, altered moods and functional limitations. Medical validation of pain cannot be performed through medical imagery in non-specific CLBP, as the relation between findings and pain is low. Following the anthropological distinction between disease, illness and sickness, patients, find themselves with "illness" (their subjective experience of suffering), but without "disease" (medical definition of the affection) or "sickness" (social construction and recognition). Lack of clear body damage explaining pain leads to an absence of social recognition as a sick person needing to be supported by the society.

Living with CLBP: a biographical disruption

Chronic symptoms can lead to a feeling of hopelessness, depression, anger and a loss of self and identity. The loss of social role, status and identity induced by chronic illness is documented in medical socio-anthropology. As shown in socio-anthropological studies on chronic illness, there is a biographical disruption when the illness appears. The CLBP patient has to manage his life accounting for pain. Self-image is altered and a feeling of self-discrepancy, i.e. a difference between ideal and perceived self, may be experienced.

Some patients feel that there are held responsible for their suffering, when physicians situate the origin of pain "in the mind" in the absence of identified body damage. Patients often consider that physicians don't admit the limitations of medicine. Persons in unexplained pain, speak of solving the riddle which they can't resign to consider as "imagined pain". They are often convinced of the concreteness of their pain, since "you can't hurt this bad and there being nothing wrong". Some complain "having been let down" in this quest and explain they had to cope on their own with their situation.

Although these studies show the importance of taking into account the lived situations and trajectory of the ill persons since the beginning of the illness, they make little articulation between these trajectories and ill persons' expectations towards caregivers. In this study the investigators assume there are strong links between these aspects. For instance, the duration of the illness, the level of disability, its impact on the quality of life, the previous recourse to other therapists and treatments necessarily produce variations in the patients' expectations towards the physiotherapists.

Research aims

The main aim of this study is to identify CLBP patients' expectations toward physiotherapy and physiotherapists. The investigators will aim at providing a qualitative insight into the factors influencing the expectations by relating them to the experience and elements of the context in which they appear. The elements accounted for will include the representation of CLBP, physiotherapy and its therapists, the illness trajectory, the socio-economic characteristics, the techniques and the perceived relationship with the physiotherapists. Expectations will be investigated at the beginning and the end of an intensive rehabilitation program to seize how this experience answers and/or modifies the patient's expectations.

Methodology

Design: individual interviews and observations

Interviews with patients and observations of the patient-physiotherapist interactions are planned.

Interviews

Individual comprehensive interviews are a common method to provide accounts of the experience of illness.

The investigators will use semi-structured interviews based on a guide of questions. Interviews will be conducted by the anthropologists of the research team. Interviews will last around 1 hour. They will take place at the ill person's home if he/she agrees.

At the beginning of the process, 4 pilot interviews and two individual sessions (observations) will be run to refine questions and procedures, as well as adjust to unplanned practical issues.

Two interviews will take place, one at the beginning of the rehabilitation program, and the second at the end. Both interviews will be conducted by the same researcher.

Observations

With an aim of a triangulation of data, the interviews will be completed with observations of the relationship between patients and physiotherapists.

The observations will take place in the back rehabilitation unit of the university hospital. Patients will follow a 3 week intensive CLBP rehabilitation program.

Focus will be put on individual therapy sessions. More specifically, the first and the last session of the program will be observed. The investigators will choose ten patients among the twenty participants using the same purposive sampling process.

These observations will be conducted by the two anthropologists in the research team. Following the observations, all members of the research team will meet for debriefing sessions, to share visions between anthropologists and physiotherapists about the meaning of the events. This will assure taking into account both socio-anthropological concepts and physiotherapists' knowledge of the field in an interdisciplinary approach.

ELIGIBILITY:
Inclusion Criteria:

* working age group (18 to 65 years old)
* have a medically confirmed non-specific chronic low-back pain

Exclusion Criteria:

* severe mental illness
* concurrent illness or co-morbidity interfering with the course of treatment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A purposive sample will be used. The investigators will aim at the recruitment of a diversified sample of patients following an intensive chronic low back pain rehabilitation program. The sample will include as many men as women, as many young than older participants (3 age groups: 18-30, 30-50, 50-65), as much variety in educational level and occupation as possible. The type of work (physical demand of employment) and career track will also be taken into account, as well as having a representation of migrants (since they are overrepresented in the back pain population58). It is estimated that data saturation should be reached with 20 participants.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2014-04; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Expectations at baseline | 2 weeks before a rehabilitation program
  Qualitative data on patient's expectations toward physiotherapy and physiotherapists issued from interviews and observations

SECONDARY OUTCOMES:
Factors influencing expectations at baseline | 2 weeks before a rehabilitation program
  Qualitative data on factors influencing expectations. This includes patient's characteristics (sex, age,..), representation of CLBP, representation of physiotherapy and physiotherapists, illness trajectory, socio-economic characteristics, treatment techniques and perceived relationship with the physiotherapists.
Factors influencing expectations at T2 | 2 weeks after a rehabilitation program
  Qualitative data on factors influencing expectations. This includes patient's characteristics (sex, age,..), representation of CLBP, representation of physiotherapy and physiotherapists, illness trajectory, socio-economic characteristics, treatment techniques, treatment outcome, intensive rehabilitation treatment experience and perceived relationship with the physiotherapists.
Expectations at T2 | 2 weeks after a rehabilitation program
  Qualitative data on patient's expectations toward physiotherapy and physiotherapists issued from interviews and observations

CONTACTS AND LOCATIONS:
Overall Officials: Claude Pichonnaz, PT, MSc, Study Director — Hautre Ecole de Santé Vaud, physiotherapy department; Rose-Anna Foley, PhD, Principal Investigator — Haute Ecole de Santé Vaud, research unit
Locations (1):
- Chuv-Unil, Lausanne, Canton of Vaud, Switzerland